CLINICAL TRIAL: NCT01937676
Title: LDH as a Biochemical Biomarker to Predict Organ Failure in the Emergency Department Setting
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Fredrik Helliksson, MD, Karolinska Institutet
Other Study IDs: K3-akuten
Record Dates: First submitted 2013-08-30; First posted 2013-09-09 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Organ Failure
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults admitted to ER: All adult patients admitted to emergency department during the study period.

SUMMARY:
The purpose of this study is evaluate if K3, a novel biomarker, sampled at arrival to the emergency department can be used to predict the development of organ failure measured as SOFA score. K3 consists of lactate dehydrogenase, albumin and magnesium combined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Admitted to emergency department, Karlstad Central Hospital, Sweden

Exclusion Criteria:

* Not in need of venous blood sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to emergency department during study period.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Development of multiple organ failure | 30 days or complete ICU stay
  Measured as SOFA score.

SECONDARY OUTCOMES:
Cardiac function | 30 days or complete ICU stay
  Is it possible to predict cardiac function with the novel biomarker K3, which consists of lactate dehydrogenase, albumin, and magnesium combined?
All cause mortality | 30 days after admission to emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Karlsson, MD, PhD, Principal Investigator — Karolinska; Jan Wernerman, MD, Prof, Study Director — Karolinska; Lars Wiklund, MD, Prof, Study Director — Uppsala University
Locations (1):
- Karlstad Central Hospital, Karlstad, Sweden